CLINICAL TRIAL: NCT06170944
Title: Effect of Remote Ischemic Preconditioning on Collaterals of Atherosclerosis Stroke (RICAS): a Prospective, Randomized, Blind Endpoint, Multicenter Study
Brief Title: Effect of Remote Ischemic Preconditioning on Collaterals of Atherosclerosis Stroke
Acronym: RICAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y(2023)169
Record Dates: First submitted 2023-12-05; First posted 2023-12-14 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic preconditioning and guideline-based treatment (Experimental): 5 cycles of cuff inflation (200mmHg for 5 minutes) and deflation (for 5 minutes), once or twice daily for 12 months.
  Interventions: Device: Remote ischemic preconditioning
- Guideline-based treatment (No Intervention): Guideline-based treatment.

INTERVENTIONS:
Device: Remote ischemic preconditioning — The patients in experiment group will receive treatment with RIC (5 cycles of cuff inflation for 5 minutes and deflation for 5 minutes to the bilateral upper limbs to 200 mmHg) for 1 year as an adjunct to guideline-based treatment.
  Arms: Remote ischemic preconditioning and guideline-based treatment

SUMMARY:
The goal of this clinical trial is to explore the influence of chronic RIC on collateral status evaluated by DSA in ischemic stroke patients with LAA etiology.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death and the third leading cause of death and disability combined in the world. The remote ischemic preconditioning (RIC) procedure is low-cost with excellent properties of safety, tolerability and feasibility in both AIS and cardiovascular diseases. In this study, we aim to explore the influence of chronic RIC on collateral status evaluated by DSA in ischemic stroke patients with LAA etiology. The RICAS study is a prospective, randomized, blind endpoint, multicenter study. Eligible patients with ischemic stroke of anterior circulation with large artery atherosclerosis etiology, poor collateral compensation, and more than 1 month of the symptom onset, are randomly assigned into the experimental group and control group with a ratio of 1:1. The patients in experiment group will receive treatment with RIC for 1 year as an adjunct to guideline-based treatment, while patients in control group only receive guideline-based treatment. The primary outcome is proportion of collateral status improvement, which is defined as an increase of ASITN/SIR score of 1 or more assessed on DSA at 12 months after randomization. The safety outcomes include RIC-related adverse events. A maximum of 300 patients (150 participants per group) are required to test the superiority hypothesis with 80% power (using a two-sided α = 0.05) to detect the 15% difference. The primary endpoint will further be stratified by age, gender, inclusion event (acute ischemic stroke ore transient ischemic stroke), tandem lesion, history of hypertension, hypercholesterolemia, diabetes mellitus, ischemic stroke, transient ischemic attack, and myocardial infarction. This study will provide the direct evidence for improvement of collateral status by chronic RIC treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age over 40 years old;
* 2. Diagnosed with ischemic stroke (including TIA and cerebral infarction), with onset time of more than 1 month;
* 3. Culprit arteries are the large arteries of the anterior circulation with atherosclerotic stenosis (≥50%) or occlusion;
* 4. ASITN/SIR collateral circulation of 0-3 based on DSA evaluation;
* 5. First onset or prior onset with no significant sequelae (mRS ≤ 2);
* 6. Those who are not expected to undergo angioplasty within 12 months (judged by the doctor or decided by patients and/or their representatives);
* 7. The availability of informed consent.

Exclusion Criteria:

* 1) Patients with severe infection or serious diseases such as liver, kidney, hematopoietic system, endocrine system, etc.;
* 2) Patients with a history of stroke and severe sequelae (mRS≥3);
* 3) arterial stenosis due to aortic dissection, moyamoya disease; Any known vasculitic disease; herpes zoster, varicella-zoster or other viral infections with vascular lesions; neurosyphilis; other intracranial infections; any intracranial artery stenosis associated with hypercytosis of cerebrospinal fluid; radiation-induced vascular lesions; myofiber dysplasia; sickle cell disease; neurofibromas; benign vascular lesions of the central nervous system; postpartum vascular disease; stenosis of the intracranial arteries due to vasospasm or thrombosm;
* 4) Uncontrolled severe hypertension (systolic pressure≥180mmHg or diastolic pressure≥110 mmHg after drug treatment) ;
* 5) Subclavian artery stenosis ≥50% or subclavian artery steal syndrome;
* 6) Patients with intracranial hemorrhage (parenchymal hemorrhage, subarachnoid hemorrhage, subdural/epidural hemorrhage) within 90 days before enrollment;
* 7) Intracranial tumor, arteriovenous malformation, or aneurysm;
* 8) Patients with severe hematologic diseases or severe coagulation abnormalities;
* 9) Retinal hemorrhage or visceral hemorrhage within 30 days;
* 10) Those who are expected to undergo major surgery (including femoral artery, cardiac, aortic or carotid artery surgery) within 30 days before enrollment or within 12 months after enrollment;
* 11) Those who have received stent implantation, angioplasty or other related medical devices for the target diseased blood vessels, or those who are expected to undergo the above treatments within 12 months after enrollment;
* 12) Any contraindication for remote ischemic adaptation: the upper limb has serious soft tissue injury, fracture or vascular injury, distal upper limb perivascular lesions, etc.
* 13) Damage and lesions in the cerebral veins;
* 14) Pregnant or lactating women;
* 15) Those who are participating in other clinical trials within 3 months;
* 16) Life expectancy is less than 1 year
* 17) Patients not suitable for this clinical studies considered by researcher

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of collateral status improvement. | 12 months
  collateral status improvement is defined as an increase of ASITN/SIR score of 1 or more assessed on DSA at 12 months after randomization.

SECONDARY OUTCOMES:
The influence of RIC to neurological functions | 12 months
  Neurological functions was determined by modified Rankin Scale score (0-42, higher scores mean a worse outcome )
Recurrence of nonfatal ischemic stroke in 12 months | 12 months
  Ischemic stroke is diagnosed based on clinical symptom and neuroimaging
Composite vascular events | 12 months
  Composite vascular events include stroke, myocardial infarction, vascular death
Influence on heart function | 12 months
  heart function is assessed by cardiac ultrasound, electrocardiogram, myocardial enzyme profile, etc
Influence on kidney function | 12 months
  kidney function is assessed by glomeruar filtration rate
RIC-related adverse events | 12 months
  include local pain, intolerance, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: Yes
Data dictionary.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: With publication.
Access Criteria: Researchers whose proposed use of the data has been approved.

REFERENCES:
- [Derived] Zhao ZA, Lv Y, Chen HS. Effect of RICAS (Remote Ischemic Preconditioning on Collaterals of Atherosclerosis Stroke): Rationale and Design. J Am Heart Assoc. 2025 Mar 18;14(6):e038570. doi: 10.1161/JAHA.124.038570. Epub 2025 Feb 19. PMID 39968799